CLINICAL TRIAL: NCT07155330
Title: High-flow Nasal Cannula Oxygenation in Sedated Endoscopy for High-risk Obstructive Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chief Physician,Researcher, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025C128
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Hypoxemia; Esophageal Cancer; Gastric Cancer (Diagnosis); Colon Cancer
Keywords: High-Flow Nasal Oxygen; Hypoxemia; Gastrointestinal Endoscopy; Sedation; obstructive sleep apnea
MeSH Terms: conditions — Hypoxia; Esophageal Neoplasms; Stomach Neoplasms; Disease; Colonic Neoplasms; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-flow nasal cannula (Experimental): Using high-flow nasal cannula oxygenation
  Interventions: Device: High-flow nasal cannula

INTERVENTIONS:
Device: High-flow nasal cannula — Using high-flow nasal cannula oxygenation

SUMMARY:
Hypoxia is the most common adverse event during propofol sedation for gastrointestinal endoscopy. The STOP-BANG questionnaire is a widely used, simple assessment tool for screening obstructive sleep apnea (OSA) risk. A STOP-Bang score ≥5 indicates high-risk OSA patients who are more prone to hypoxia during sedated endoscopy. Our team's preliminary clinical research found that High-Flow Nasal Cannula (HFNC) may reduce hypoxemia risk, but there are limited dedicated studies focusing specifically on high-risk OSA patients, with controversial results. This study aims to investigate whether HFNC can reduce the incidence of hypoxia during sedated gastrointestinal endoscopy in high-risk obstructive sleep apnea patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* STOP-Bang score ≥5.
* Scheduled for sedated gastrointestinal endoscopy (gastroscopy, colonoscopy, or combined gastroscopy + colonoscopy).
* The estimated duration of the procedure does not exceed 45 minutes.
* Patients have signed the informed consent form.

Exclusion Criteria:

* Coagulation disorders or bleeding tendency (e.g., oral/nasal bleeding risk, mucosal injury, space-occupying obstructions).
* Active upper respiratory tract infection (oral, nasal, or pharyngeal), or fever (core temperature >37.5°C).
* Chronic obstructive pulmonary disease or other acute/chronic pulmonary diseases requiring long-term or intermittent oxygen therapy, or preoperative SpO₂ ≤ 92% on room air.
* Severe organ dysfunction, including: Cardiac insufficiency (<4 METs), Severe renal insufficiency (requiring dialysis), Diagnosed severe hepatic insufficiency, Increased intracranial pressure, ASA physical status ≥ IV.
* Confirmed pregnancy or current breastfeeding.
* Known allergy to sedatives (e.g., propofol) or medical adhesives.
* Multiple traumatic injuries.
* Current participation in another clinical trial.
* Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO2 < 95%
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No